CLINICAL TRIAL: NCT03468920
Title: Comparison of Outcomes When Patients Receive Preoperative IV Acetaminophen Versus Preoperative Oral Acetaminophen
Brief Title: Preoperative IV Versus Oral Acetaminophen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Rachel Baker, Nurse Researcher, TriHealth Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-114
Record Dates: First submitted 2018-03-01; First posted 2018-03-19 (Actual); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study will use a randomized, double-blind, placebo controlled design with two arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only pharmacy staff will have randomization scheme and be aware of whether patient received oral Acetaminophen with IV placebo OR if the patient received IV Acetaminophen with oral placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: IV Acetaminophen group (Experimental): Patients randomized to Arm 1 will receive IV Acetaminophen 1000mg in 100mL NS once and a PO placebo pill preoperatively
  Interventions: Drug: IV Acetaminophen; Drug: PO Placebo
- Arm 2: PO Acetaminophen group (Active Comparator): Patients randomized to Arm 2 will receive IV normal saline 100mL once and Acetaminophen 1000 mg PO once preoperatively
  Interventions: Drug: PO Acetaminophen; Drug: IV Solution Placebo

INTERVENTIONS:
Drug: IV Acetaminophen — IV Acetaminophen 1000mg in 100mL normal saline once pre-operatively
  Other Names: Tylenol
  Arms: Arm 1: IV Acetaminophen group
Drug: PO Acetaminophen — Acetaminophen PO 1000mg once pre-operatively
  Other Names: Tylenol
  Arms: Arm 2: PO Acetaminophen group
Drug: PO Placebo — PO placebo capsule compounded to match PO Acetaminophen capsule
  Arms: Arm 1: IV Acetaminophen group
Drug: IV Solution Placebo — This will serve as the placebo for the IV Acetaminophen intervention
  Other Names: IV Normal Saline
  Arms: Arm 2: PO Acetaminophen group

SUMMARY:
The current study proposes to examine whether there is a significant difference in patient outcomes related to the administration route of preoperative Acetaminophen. Specifically, the study will compare outcomes of surgical patients who receive IV Acetaminophen with surgical patients who receive oral Acetaminophen.

DETAILED DESCRIPTION:
This study will use a randomized, double-blind, controlled design with two arms:

Arm 1: Scheduled IV Acetaminophen and PO placebo provided preoperatively Arm 2: Scheduled PO Acetaminophen and IV placebo provided preoperatively

120 patients will be randomized 1:1 into Arm 1 or Arm 2. All other care, except route of preoperative Acetaminophen, will follow standard care procedures. The following outcome measures will be collected: postoperative pain, postoperative opioid medication administration, postoperative nausea and vomiting, occurrence of respiratory depression postoperatively, occurrence of administration of reversal agent postoperatively, length of stay in recovery room, patient satisfaction with pain control.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Admitted to Bethesda Butler Main Perioperative Services for an outpatient surgical procedure performed under general anesthesia

Exclusion Criteria:

* Allergy to Acetaminophen
* Lactose intolerance or lactose allergy (placebo capsules contain lactose)
* Hepatic disease
* Having taken a product containing acetaminophen within 6 hours of scheduled surgery time
* Pregnant
* Weight less than 50kg
* Opioid addiction - admits to current opioid addiction and/or substance abuse disorder, and/or currently in treatment for opioid addiction or substance abuse
* Emergent or on-call procedures
* Inpatient surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TriHealth, Bethesda Butler Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: IV Acetaminophen Group | Arm 2: PO Acetaminophen Group
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: IV Acetaminophen Group | Arm 2: PO Acetaminophen Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.37 (15.82) | 46.28 (16.84) | 45.83 (16.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 23 | 25 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Pain
Description: Pain measured from 0 (no pain) to 10 (worst pain)
Time Frame: through study visit, less than 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: IV Acetaminophen Group | Arm 2: PO Acetaminophen Group
Number analyzed (Participants) | 60 | 60
score on a scale | 4.12 (3.092) | 4.37 (3.226)

2. Secondary Outcome: Number of Participants Who Received Opioid Administration in PACU
Description: Number of Participants who Received Opioid Administration in PACU
Time Frame: through study visit, less than 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IV Acetaminophen Group | Arm 2: PO Acetaminophen Group
Number analyzed (Participants) | 60 | 60
Participants | 31 | 34

3. Secondary Outcome: Number of Participants Who Experienced Postoperative Nausea and Vomiting
Description: Did patient experience negative effects of pain medication (postoperative nausea and vomiting)
Time Frame: through study visit, less than 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: IV Acetaminophen Group | Arm 2: PO Acetaminophen Group
Number analyzed (Participants) | 60 | 60
Participants | 8 | 6

4. Secondary Outcome: Length of Stay
Description: Minutes from entering PACU to end of Phase II
Time Frame: through study visit, less than 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1: IV Acetaminophen Group | Arm 2: PO Acetaminophen Group
Number analyzed (Participants) | 60 | 60
minutes | 88.25 (26.651) | 92.88 (29.911)

5. Secondary Outcome: Patient Satisfaction
Description: Patient reported satisfaction with pain control on a scale of 1 (extremely unsatisfied) to 10 (extremely satisfied)
Time Frame: up to 2 days after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: IV Acetaminophen Group | Arm 2: PO Acetaminophen Group
Number analyzed (Participants) | 60 | 60
score on a scale | 9.45 (0.950) | 9.77 (0.528)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Arm 1: IV Acetaminophen Group | Arm 2: PO Acetaminophen Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03468920/Prot_SAP_000.pdf